CLINICAL TRIAL: NCT02836015
Title: Shared Medical Visits for Spanish-speaking Patients With Type 2 Diabetes
Acronym: SMV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0146-16-EP
Record Dates: First submitted 2016-05-23; First posted 2016-07-18 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Shared Medical Visits; Spanish-speaking
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shared Medical Visit Groups (Experimental): All patients will be enrolled in the experimental group and will be involved in shared medical visits.
  Interventions: Behavioral: Shared Medical Visit

INTERVENTIONS:
Behavioral: Shared Medical Visit — The Shared Medical Visits are a replacement for standard diabetic visits with PCP, and will occur completely in Spanish, the patients' preferred primary language. An interdisciplinary group including behavioral health, social work, pharmacy, MD, and diabetic educator will be involved in the visit. The focal point of the meeting is a 30 minute session in which all members are seated around a large table in the Midtown SMV area and each patient's blood sugars, labs, and medications are discussed in front of the entire group. Pertinent labs and vaccines are drawn/administered.
  Other Names: SMV

SUMMARY:
The investigators seek to apply a shared medical visit model and interdisciplinary approach to Spanish-speaking patients. The investigators will evaluate the patient's hemoglobin A1c as a marker of glycemic control and evaluate their mood with PHQ screening tools. The investigators seek to improve diabetes care for this group of underserved patients. Potential participants will be selected from the UNMC diabetes registry. Eligibility criteria includes adult patients over the age of eighteen years old with Type 2 diabetes, HgbA1c greater than 8%, whose preferred language is Spanish. Exclusion criteria include pregnancy, residency at a nursing home or other facility, substance abuse, and physician recommendation that study is not appropriate for the patient.

DETAILED DESCRIPTION:
Type 2 diabetes is an expanding epidemic, which is particularly pervasive in the Hispanic community. In 2014, the CDC reported that 21.9 million adults have been diagnosed with diabetes, a number which has nearly quadrupled since 1980.

Diabetes is a particularly challenging chronic disease due to the need for self-management. This research study plans to explore how shared medical visits with Spanish-speaking patients with diabetes can improve their control of diabetes, develop self-management behaviors, and enhance overall perspective of having a chronic disease.

The investigators will model this project after an ongoing with English speakers and they have demonstrated improvements in hemoglobin A1c levels and quality of life, and will now apply this model to Spanish-speaking patients.

Eligibility and exclusion criteria are detailed in the brief summary. Eligible participants will be recruited for the study through use of phone call in Spanish, letter writing in Spanish, word of mouth, and direct referral from their providers throughout UNMC. Once the list of potential subjects is compiled, those patients will be contacted and the details of the study will be explained in Spanish. All the participating staff in the study speak Spanish. The participants, at any time, can withdraw from the study.

Participants will receive education in diabetes health and lifestyle education. This will be a quantitative study using pre- and post-intervention measures to evaluate the outcomes of HgbA1c levels, scores on the validated 2-item and 9-item Patient Health Questionnaires (PHQ-2 and PHQ-9), and questionnaire which measures improvements in self-management behaviors.

Researchers will to follow-up with the participants in the week following the visit to discuss lab results. At the end of the study, researcher will send a detailed letter to the patient's primary care provider regarding progress and management in shared medical visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of eighteen years old with Type 2 diabetes
* HgbA1c greater than 8%
* Preferred language is Spanish

Exclusion Criteria:

* Pregnancy
* Residency at a nursing home or other facility
* Substance abuse
* Physician recommendation that study is not appropriate for the patient

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Every three months, up to 1 year
  Every 3 months we will measure hemoglobin A1c to assess for improvement in glycemic control.

SECONDARY OUTCOMES:
Improvement in self care behaviors | Every three months, up to 1 year
  See improvement in self care behaviors as defined by American Association of Diabetes Educators1: healthy eating, being active, monitoring, taking medication, problem solving, reducing risks, and healthy coping
Barriers to care for Spanish-speaking patients with diabetes | Every 3 months, up to 1 year
  Identify barriers to care for Spanish-speaking patients with diabetes, which are specific to this minority group, in order to improve care of this specific population.
Screening for complications of diabetes | Once annually, up to 1 year
  Urine microalbumin/creatinine ratio, low density lipoprotein, yearly dilated eye exam, yearly flu shot, and yearly diabetic foot exam.
PHQ-2 and PHQ-0 Depression screening tool | Every three months, up to 1 year
  Evaluate change in the overall mood of patients with diabetes, as measured by reduced scores on the validated depression screening assessments. Each patient will always be administered the PHQ-2, a 2 question survey, and if they screen positive for depression on that they will be administered a PHQ-9, 9 question depression screening tool.
Blood pressure | Every 3 months, up to 1 year
  Assessment of blood pressure at each visit, with goal for improvement in blood pressure control.
BMI | Every 3 months, up to 1 year
  Participants will have height and weight measured at each visit which allows for calculation of BMI

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Eiland, MD, Principal Investigator — University of Nebraska
Locations (1):
- Nebraska Medicine, Midtown Health Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edelman D, Gierisch JM, McDuffie JR, Oddone E, Williams JW Jr. Shared medical appointments for patients with diabetes mellitus: a systematic review. J Gen Intern Med. 2015 Jan;30(1):99-106. doi: 10.1007/s11606-014-2978-7. Epub 2014 Aug 9. PMID 25107290
- [Background] Trento M, Passera P, Tomalino M, Bajardi M, Pomero F, Allione A, Vaccari P, Molinatti GM, Porta M. Group visits improve metabolic control in type 2 diabetes: a 2-year follow-up. Diabetes Care. 2001 Jun;24(6):995-1000. doi: 10.2337/diacare.24.6.995. PMID 11375359
- [Background] McCloskey J, Flenniken D. Overcoming cultural barriers to diabetes control: a qualitative study of southwestern New Mexico Hispanics. J Cult Divers. 2010 Fall;17(3):110-5. PMID 20860336
- [Background] Ramal E, Petersen AB, Ingram KM, Champlin AM. Factors that influence diabetes self-management in Hispanics living in low socioeconomic neighborhoods in San Bernardino, California. J Immigr Minor Health. 2012 Dec;14(6):1090-6. doi: 10.1007/s10903-012-9601-y. PMID 22427108
- [Background] Pyatak EA, Florindez D, Peters AL, Weigensberg MJ. "We are all gonna get diabetic these days": the impact of a living legacy of type 2 diabetes on Hispanic young adults' diabetes care. Diabetes Educ. 2014 Sep-Oct;40(5):648-58. doi: 10.1177/0145721714535994. Epub 2014 May 27. PMID 24867918
- [Background] Ell K, Katon W, Xie B, Lee PJ, Kapetanovic S, Guterman J, Chou CP. Collaborative care management of major depression among low-income, predominantly Hispanic subjects with diabetes: a randomized controlled trial. Diabetes Care. 2010 Apr;33(4):706-13. doi: 10.2337/dc09-1711. Epub 2010 Jan 22. PMID 20097780
- [Result] Bohn J, Burrowes N, Pinkston L, Riddett M, Chalmers S. Diabetes care for Hispanic patients: honoring culture while promoting glycemic control. Adv Nurse Pract. 2010 Jan;18(1):46-8. No abstract available. PMID 20128205
- [Result] Jaber R, Braksmajer A, Trilling JS. Group visits: a qualitative review of current research. J Am Board Fam Med. 2006 May-Jun;19(3):276-90. doi: 10.3122/jabfm.19.3.276. PMID 16672681
- [Result] Gutierrez N, Gimple NE, Dallo FJ, Foster BM, Ohagi EJ. Shared medical appointments in a residency clinic: an exploratory study among Hispanics with diabetes. Am J Manag Care. 2011 Jun 1;17(6 Spec No.):e212-4. PMID 21756014
- See also: Diabetes Initiative: a National Program of The Robert Wood Johnson Foundation — http://www.diabetesinitiative.org